CLINICAL TRIAL: NCT02331238
Title: Cluster-Randomized Trial of a Middle School Coach Gender Violence Prevention Program
Brief Title: Trial of a Middle School Coach Gender Violence Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elizabeth Miller, Chief, Division of Adolescent and Young Adult Medicine, Children's Hospital, University of Pittsburgh Medical Center, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO14020618
Record Dates: First submitted 2015-01-01; First posted 2015-01-06 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Violence; Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control School (No Intervention): Control schools (where the coaches do not receive the "Coaching Boys into Men" training until following academic year ;wait list control)
- Intervention School (Experimental): Intervention schools (where coaches receive the Coaching Boys into Men training at start of each sports season).
  "Coaching Boys into Men" program consists of 60 minute training for high school coaches led by a violence prevention advocate to introduce coaches to the rational for Coaching Boys into Men and the Coaching Boys into Men Coaches Kit. The coaches use this Coaching Boys into Men toolkit to provide weekly discussions with their athletes (generally 10-15 minute mini-sessions) throughout their athletic season (11 weeks). Discussion topics include how to prevent disrespectful and harmful behaviors towards women and girls and how to promote healthy choices and relationships among youth.
  Interventions: Behavioral: "Coaching Boys into Men" program

INTERVENTIONS:
Behavioral: "Coaching Boys into Men" program — "Coaching Boys into Men" program consists of 60 minute training for high school coaches led by a violence prevention advocate to introduce coaches to the rational for Coaching Boys into Men and the Coaching Boys into Men Coaches Kit. The coaches use this Coaching Boys into Men toolkit to provide weekly discussions with their athletes (generally 10-15 minute mini-sessions) throughout their athletic season (11 weeks). Discussion topics include how to prevent disrespectful and harmful behaviors towards women and girls and how to promote healthy choices and relationships among youth.
  Arms: Intervention School

SUMMARY:
This cluster-randomized school-based study will examine the effectiveness of a program for the primary prevention of perpetration of teen dating violence and sexual violence among middle school male athletes. Engaging men and boys in preventing violence against women and girls is recognized by major global health organizations as a critical public health strategy. "Coaching Boys into Men" is a theory- and evidence based program intended to alter gender norms that foster teen dating violence/sexual violence perpetration, promote bystander intervention, and reduce teen dating violence/sexual violence perpetration. Coaches receive a 60-minute training and biweekly check-in from a violence prevention advocate to administer the intervention to their athletes via 12 mini-lessons conducted weekly throughout a sport season. In a randomized trial of program effectiveness among high school athletes (Centers for Disease Control and Prevention CE001561-01, PI Miller), male athletes receiving the program demonstrated increased positive bystander intervention behaviors and less verbal abuse perpetration compared to controls. This project seeks to test the effectiveness of this program with younger male athletes in grades 6-8.The innovations are three-fold: (1) testing the efficacy of a novel teen dating violence/sexual violence prevention program for middle school male athletes; (2) training athletic coaches in Teen Dating Violence/Sexual Violence prevention thus implementing primary prevention that does not rely on teachers or classroom time; and (3) integrating the goal of changing gender norms with the technique of a bystander intervention approach to reduce teen dating violence/sexual violence prevention. The experimental design involves a 2-armed cluster randomized- controlled trial in 41 middle schools (38 clusters) in Pennsylvania. Schools will be randomly assigned to either intervention or control (standard coaching) condition. Coaches in intervention schools will receive Coaching Boys into Men training. Baseline surveys will be collected for all intervention and control site athletes entering grades 6-8 at the start of each sports seasons across Year 1 (Time 1; N= 973 athletes). Follow up surveys will be collected at the end of each sports season (Time 2). All participating athletes will be re-surveyed 12 months after baseline (Time 3).

ELIGIBILITY:
Inclusion Criteria:

School eligibility:

Urban and suburban middle schools in the Pittsburgh, PA region with athletics program

Athlete eligibility:

Ages 11-14 (grades 6-8), student at a participating middle school, participating in an athletic program led by coach participating in the research study

Exclusion Criteria:

School Eligibility:

Middle schools not in the Pittsburgh area

Athlete eligibility:

Outside age range, not participating on a sports team at the middle school in which they are enrolled

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 973 (Actual)
Dates: Start 2015-03; Primary Completion 2017-11-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in Positive Bystander Behavior from Baseline to Follow Up | 3 months and 12 months
  Assessment of past 3 month positive bystander behavior in athletes when witnessing disrespectful and harmful behavior among peers comparing baseline and follow up summary scores. Athletes report if they have witnessed peers' abusive behaviors in the past 3 months and if witnessed, how they responded (whether they intervened to interrupt the behavior)

SECONDARY OUTCOMES:
Change in Recognition of Abusive Behavior from Baseline to Follow Up | 3 months and 12 months
  Recognition of disrespectful and harmful behaviors against girls as abusive comparing baseline and follow up mean scores on the recognition of abusive behavior scale.
Change in Gender Equitable Attitudes Scale from Baseline to Follow Up | 3 months and 12 months
  Assessment of gender-equitable attitudes comparing baseline and follow up mean scores on the gender attitudes scale
Change in Intentions to Intervene from Baseline to Follow Up | 3 months and 12 months
  Proclivity to intervene when witnessing disrespectful and harmful behaviors among peers comparing baseline and follow up mean scores on a scale assessing likelihood of trying to stop disrespectful behaviors among peers.
Change in self-reported recent (past 3 month) perpetration of Teen Dating Violence/Sexual Violence at 12 months | 12 Months
  Assessment of Teen Dating Violence/Sexual Violence perpetration comparing baseline summary score with follow up 12 month summary score (whether participants have perpetrated acts of Teen Dating Violence or Sexual Violence towards anyone)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Miller E, Tancredi DJ, McCauley HL, Decker MR, Virata MC, Anderson HA, Stetkevich N, Brown EW, Moideen F, Silverman JG. "Coaching boys into men": a cluster-randomized controlled trial of a dating violence prevention program. J Adolesc Health. 2012 Nov;51(5):431-8. doi: 10.1016/j.jadohealth.2012.01.018. Epub 2012 Mar 25. PMID 23084163
- [Background] Miller E, Tancredi DJ, McCauley HL, Decker MR, Virata MCD, Anderson HA, O'Connor B, Silverman JG. One-year follow-up of a coach-delivered dating violence prevention program: a cluster randomized controlled trial. Am J Prev Med. 2013 Jul;45(1):108-112. doi: 10.1016/j.amepre.2013.03.007. PMID 23790995
- [Derived] Jones KA, Tancredi DJ, Abebe KZ, Paglisotti T, Miller E. Cases of Sexual Assault Prevented in an Athletic Coach-Delivered Gender Violence Prevention Program. Prev Sci. 2021 May;22(4):504-508. doi: 10.1007/s11121-021-01210-1. Epub 2021 Jan 22. PMID 33481150
- [Derived] Miller E, Jones KA, Ripper L, Paglisotti T, Mulbah P, Abebe KZ. An Athletic Coach-Delivered Middle School Gender Violence Prevention Program: A Cluster Randomized Clinical Trial. JAMA Pediatr. 2020 Mar 1;174(3):241-249. doi: 10.1001/jamapediatrics.2019.5217. PMID 31930358
- [Derived] Abebe KZ, Jones KA, Ciaravino S, Ripper L, Paglisotti T, Morrow SE, Grafals M, Van Dusen C, Miller E. A cluster-randomized trial of a middle school gender violence prevention program: Design, rationale, and sample characteristics. Contemp Clin Trials. 2017 Nov;62:11-20. doi: 10.1016/j.cct.2017.08.007. Epub 2017 Aug 15. PMID 28821469